CLINICAL TRIAL: NCT00102011
Title: Colonoscopy Screening Trial
Brief Title: Colonoscopy or Fecal Occult Blood Test in Screening Healthy Participants for Colorectal Cancer
Acronym: 00-046
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 00-046; MSKCC-00046A; UMN-2003NT062
Record Dates: First submitted 2005-01-18; First posted 2005-01-19 (Estimated); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Colorectal Cancer
Keywords: colon cancer; rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Occult Blood

ARMS (4):
- Study I- Arm I (Experimental): Participants undergo baseline screening colonoscopy
  Interventions: Procedure: screening colonoscopy
- Study I- Arm II (Other): Participants receive standard care
  Interventions: Procedure: fecal occult blood test; Procedure: standard follow-up care
- Study II- Arm I (Experimental): Participants undergo baseline screening colonoscopy. Participants are given individualized recommendations for further surveillance based on the results of the colonoscopy.
  Interventions: Procedure: screening colonoscopy
- Study II- Arm II (Active Comparator): Participants undergo a baseline fecal occult blood test (FOBT). Participants are given individualized recommendations for further surveillance based on the results of the FOBT. Participants with negative baseline FOBT undergo FOBT annually for up to 4 years in the absence of a positive FOBT.
  Interventions: Procedure: annual screening; Procedure: fecal occult blood test

INTERVENTIONS:
Procedure: annual screening — Participants with negative baseline FOBT undergo FOBT annually for up to 4 years in the absence of a positive FOBT
  Arms: Study II- Arm II
Procedure: fecal occult blood test — Participants undergo a baseline fecal occult blood test (FOBT)
  Arms: Study I- Arm II; Study II- Arm II
Procedure: screening colonoscopy — Patients undergo baseline screening colonoscopy
  Arms: Study I- Arm I; Study II- Arm I
Procedure: standard follow-up care — Standard care
  Arms: Study I- Arm II

SUMMARY:
RATIONALE: Screening tests, such as colonoscopy and fecal occult blood test, may help doctors find tumor cells early and plan better treatment for colorectal cancer.

PURPOSE: This randomized phase III trial is studying colonoscopy to see how well it works compared to fecal occult blood test in screening healthy participants for colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the neoplastic outcome of participants at average risk for colorectal cancer who undergo colonoscopy vs annual fecal occult blood tests.
* Compare the endoscopic and clinical resources required for these screening methods in these participants.
* Compare the benefit-to-harm ratio in participants undergoing these screening methods.
* Determine the level of participation of participants undergoing these screening methods.

OUTLINE: This is a randomized, two-part, multicenter study.

Participants are asked whether they are interested in participating in a randomized controlled trial of colorectal cancer screening.

* Screening colonoscopy feasibility study I (accrual completed as of 12/14/2004): Participants who are interested in participating in a screening trial are randomized to 1 of 2 screening arms.

  * Arm I: Participants undergo baseline screening colonoscopy.
  * Arm II: Participants receive standard care.
* Screening colonoscopy feasibility study II: Participants who are interested in participating in a screening trial are randomized to 1 of 2 screening arms.

  * Arm I: Participants undergo baseline screening colonoscopy. Participants are given individualized recommendations for further surveillance based on the results of the colonoscopy.
  * Arm II: Participants undergo a baseline fecal occult blood test (FOBT). Participants are given individualized recommendations for further surveillance based on the results of the FOBT. Participants with negative baseline FOBT undergo FOBT annually for up to 4 years in the absence of a positive FOBT.

All participants are followed annually for up to 4 years.

PROJECTED ACCRUAL: A total of 1,402 participants (701 per screening arm) have been accrued for feasibility study I within 3 years (accrual completed as of 12/14/2004). An additional 3,550 participants (1,775 per screening arm) will be accrued for feasibility study II within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Healthy participants at average risk for developing colorectal cancer
* No history of colorectal cancer
* No history of familial adenomatous polyposis
* More than 5 years since prior flexible sigmoidoscopy
* No prior colonoscopy

PATIENT CHARACTERISTICS:

Age

* 50 to 69 (40 to 69 at the Louisiana State University participating site)

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Cardiovascular

* No myocardial infarction within the past year
* No congestive heart failure

Pulmonary

* No chronic obstructive pulmonary disease

Gastrointestinal

* No history of ulcerative colitis
* No history of Crohn's disease
* No history of inflammatory bowel disease

Other

* No serious comorbid condition
* No consumption of red meat within 3 days prior to and during FOBT (feasibility study II, arm II only)

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No concurrent chemotherapy other than for nonmelanoma skin cancer

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No vitamin C consumption > 250 mg within 3 days prior to and during fecal occult blood testing (FOBT) (feasibility study II arm II only)
* No nonsteroidal anti-inflammatory drugs within 7 days prior to and during FOBT (feasibility study II, arm II only)
* No concurrent anticoagulants
* No concurrent anticancer therapy except for treatment of nonmelanoma skin cancer

Ages: 40 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4952 (Estimated)
Dates: Start 2000-05; Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Neoplastic findings as assessed by screening colonoscopy vs annual fecal occult blood test (FOBT)-directed colonoscopy | 5 years
Burden on endoscopic and clinical resources | 5 years
Harms associated with screening colonoscopy vs annual FOBT-directed colonoscopy | 5 years
Benefit-to-harm ration for screening colonoscopy vs annual FOBT-directed colonoscopy | 5 years
Level of participation in screening with FOBT-directed colonoscopy vs a single colonoscopy | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ann Zauber, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - Feist-Weiller Cancer Center at Louisiana State University Health Sciences, Shreveport, Louisiana
  - Masonic Cancer Center at University of Minnesota (Data collection only), Minneapolis, Minnesota
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Kaiser Permanente Washington Health Research Institute (Data collection only), Seattle, Washington

REFERENCES:
- [Background] Shaukat A, Church TR, Shanley R, Kauff ND, O'Brien MJ, Mills GM, Jordan PA, Allen JA, Kim A, Feld AD, Zauber AG, Winawer SJ. Development and validation of a clinical score for predicting risk of adenoma at screening colonoscopy. Cancer Epidemiol Biomarkers Prev. 2015 Jun;24(6):913-20. doi: 10.1158/1055-9965.EPI-14-1321. Epub 2015 Mar 23. PMID 25800242
- [Background] Mendelsohn RB, Winawer SJ, Jammula A, Mills G, Jordan P, O'Brien MJ, Close GM, Dorfman M, Church TR, Mandelson MT, Allen J, Feld A, Kauff ND, Morgan GA, Kumar JMR, Serrano V, Bayuga-Miller S, Fischer SE, Kuk D, Zauber AG. Adenoma Prevalence in Blacks and Whites Having Equal Adherence To Screening Colonoscopy: The National Colonoscopy Study. Clin Gastroenterol Hepatol. 2017 Sep;15(9):1469-1470. doi: 10.1016/j.cgh.2017.04.014. Epub 2017 Apr 15. No abstract available. PMID 28419856
- [Derived] Zauber AG, Winawer SJ, O'Brien MJ, Mills GM, Allen JI, Feld AD, Jordan PA, Fleisher M, Orlow I, Meester RGS, Lansdorp-Vogelaar I, Rutter CM, Knudsen AB, Mandelson M, Shaukat A, Mendelsohn RB, Hahn AI, Lobaugh SM, Soto Palmer B, Serrano V, Kumar JR, Fischer SE, Chen JC, Bayuga-Miller S, Kuk D, O'Connell K, Church TR. Randomized Trial of Facilitated Adherence to Screening Colonoscopy vs Sequential Fecal-Based Blood Test. Gastroenterology. 2023 Jul;165(1):252-266. doi: 10.1053/j.gastro.2023.03.206. Epub 2023 Mar 21. PMID 36948424
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm